CLINICAL TRIAL: NCT00632645
Title: Neuroleptic and Huntington Disease. Comparison of : Olanzapine, la Tetrabenazine and Tiapride. A Multicentric, Randomised, Controlled Study.
Brief Title: Neuroleptic and Huntington Disease Comparison of : Olanzapine, la Tetrabenazine and Tiapride
Acronym: NEUROHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P060211
Record Dates: First submitted 2008-02-29; First posted 2008-03-11 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Huntington Disease
Keywords: Huntington; Neuroleptic; Unified Huntington Disease Rating Scale (UHDRS); Independence Scale; Neuroleptic Prescription required
MeSH Terms: conditions — Huntington Disease | interventions — Olanzapine; Tetrabenazine; Tiapride Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Olanzapine Mylan
  Interventions: Drug: Olanzapine
- 2 (Active Comparator): Xenazine
  Interventions: Drug: Xenazine
- 3 (Active Comparator): Tiapridal
  Interventions: Drug: Tiapridal

INTERVENTIONS:
Drug: Olanzapine — Olanzapine Mylan oral dispersible form 5 to 10 mg / 2,5 à 20 mg per day
  Other Names: Olanzapine Mylan
  Arms: 1
Drug: Xenazine — Xenazine (tetrabenazine) tabs of 25mg , from 25 mg to 200 mg
  Other Names: tetrabenazine
  Arms: 2
Drug: Tiapridal — Tiapridal (Tiapride), tabs 100 mg / from 300 to 800 mg per day
  Other Names: tiapride
  Arms: 3

SUMMARY:
Huntington's disease (HD) is autosomal dominant neurodegenerative disease, starting in average (with high variability) in the fourth decade. The disease progression is classically characterized by a cognitive deterioration (cortical-frontal dementia), motor disorders (associating chorea, dystonia and bradykinesia), psychiatric disturbances (combining depression and irritability) and metabolic disorder (cachexia). The disease is fatal within 15 to 20 years in most patients. HD has no cure. Neuroleptics are the main drug used and the only to demonstrate its efficacy on chorea in clinical trials. But neuroleptics have also beneficial and adverse effects on other disease characteristics (motor, psychiatric, cognitive or metabolic). Their profile between beneficial and adverse effects could be different according the neuroleptics and their classification. The aim of this study is to compare beneficial and adverse effects of 3 different neuroleptics in HD.

DETAILED DESCRIPTION:
We proposed a randomized controlled trial, including 180 patients, in 3 groups: Olanzapine, Tetrabenazine and Tiapride, followed during 12 months. These treatments have been selected according their profile and their frequency of use.

The principal criteria is the Independence scale, one of the functional scales of the Unified Huntington's Disease Rating Scale, the only validated scale in HD.

Secondary criteria will assess motor,functional, psychiatric and cognitive functions, metabolic parameters, tolerance and cost.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic disease with motor, behavioural and/or psychiatric disorder required medical treatment.
2. HD diagnosed with abnormal number of CAG repeats: 38 ≤ nucleotide expansion (CAG) (amendment n°5 suppressed the limit ≤ 48)
3. Neuroleptic Prescription required.
4. Age ≥ 18 (amendment n°5 suppressed the limit ≤ 65 years old)
5. Patient gave its written consent
6. Realization of medical examination and a Electroencephalogram

Exclusion Criteria:

1. Severe cognitive impairment or neuropsychiatric troubles.
2. Existing diabetes.
3. Neuroleptic prescription forbidden according to the neurologist decision.
4. Current participation to another clinical trial.
5. No drug compliance to previous treatment.
6. No national health insurance affiliation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
the Independence scale | at 12 month

SECONDARY OUTCOMES:
motor scale | at 3, 6, 9 and 12 month
Psychiatric scale | at 3, 6, 9 and 12 month
cognitive function scale | at 3, 6, 9 and 12 month
metabolic parameters | at 3, 6, 9 and 12 month
tolerance | at 3, 6, 9 and 12 month
cost | at 3, 6, 9 and 12 month
Function scale (TFC and Functionnal Appreciation Scale) | at 3, 6, 9 and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Catherine BACHOUD LEVI, PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- CHU Henri Mondor, Créteil, France